CLINICAL TRIAL: NCT05611970
Title: Pippa Fitness Pessary Device Effectiveness and Safety Study
Brief Title: Pippa Pessary Study (Clinical Trial)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Management decision
Sponsor: Liv Labs Inc. (Industry)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LL101; R44HD105574-02 (NIH)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; SUI; pelvic floor dysfunction
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Pessaries

STUDY DESIGN:
Intervention Model Description: Interventional multi-clinic study where each participant serves as her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): Each study participant serves as her own control.
  Interventions: Device: Vaginal pessary

INTERVENTIONS:
Device: Vaginal pessary — A reusable vaginal pessary for stress urinary incontinence

SUMMARY:
This is an open label, interventional, single arm, multi-clinic study where each adult female participant with stress urinary incontinence (SUI) serves as her own control (vaginal pessary use vs. no vaginal pessary).

DETAILED DESCRIPTION:
The overall objectives of this clinical study are to demonstrate the effectiveness and safety of the Pippa Fitness Pessary (device) when self-administered and used in a home environment. Specifically, this study will evaluate the effectiveness of the Pippa Fitness Pessary by assessing reduction in urine leakage in up to 90 women with Stress Urinary Incontinence.

Effectiveness will be assessed by percentage reduction in 1-hour pad weight gain, reduction of stress urinary incontinence episodes per day, and a quality-of-life questionnaire. The safety of the Pippa Fitness Pessary will be evaluated by assessing all adverse events, including the results of urinalysis and vaginal examination.

ELIGIBILITY:
Inclusion Criteria:

* Female, ≥18 years of age
* Diagnosed with SUI by a physician using a cough stress test (positive test)
* Confirmed Pippa Fitness Pessary fit in clinic by a physician or qualified clinician (e.g., Nurse Practitioner, Registered Nurse)
* Have a >3 month history of experiencing more than 3 episodes of SUI per week
* English literacy sufficient to understand the nature of the study and sufficient to read and understand the informed consent form
* Provision of a signed and dated informed consent form
* Willingness to use the Pippa Fitness Pessary during the study and comply with study procedures
* Willingness to forego use of any vaginal insert (e.g.: vaginal pessaries, bladder supports, estrogen rings, tampons, and menstrual cups) while the Pippa Fitness Pessary is in place
* Willingness to cease use of any other form of urinary incontinence treatment for the duration of the study
* Willingness and ability to interact with study staff by email, phone, text message and video conferencing software throughout study

Exclusion Criteria:

* Known urethral stricture, bladder neck contracture, spastic bladder, vesicoureteral reflux, bladder stones, and/or bladder tumors
* Concurrent bladder specific medications (including beta agonists or anticholinergics) that affect urination and the use of any other prescription medication and/or over-the-counter medication and/or dietary supplements (including herbal supplements and those taken as teas) that affect urination, except in those instances where they are medically necessary and can be actively supported at a stable dosage throughout the active study period
* Known prolapse beyond hymen or any POP-Q point > 0
* Known hypersensitivity to silicone rubber
* Pelvic floor surgery including anterior bladder repair and urethral slings
* Vaginal, perineal, or uterine surgery, or abortion (spontaneous or induced) within the past 3 months
* Any injectable treatments, or prior surgeries for incontinence
* Class III Obesity (BMI > 40.0 kg/m2)
* Currently suffering from urinary tract or vaginal infection
* Pregnant or planning to become pregnant within 3 months, or within 3 months postpartum
* History of Toxic Shock Syndrome or consistent symptoms
* Previously diagnosed with urge-predominant or mixed predominant urinary incontinence, functional incontinence, incontinence due to a central or spinal cord neurological condition (such as multiple sclerosis, neurogenic bladder, Parkinson's, spina bifida), insensate incontinence, or overflow incontinence
* Screening laboratory values outside the reference range considered significant by the investigator which might impact the safety of the participant or outcome of the study
* Unsuccessful fit assessment during screening
* Any other reason the investigator decides the potential participant should not participate in the study
* Self-reported difficulty emptying bladder
* Difficulty inserting or wearing an intra-vaginal device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women
Enrollment: 7 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Responder rate of success in reduction of urine leakage with intervention | 24 days
  A responder will be defined as having >50% reduction in pad weight gain for the 1-hour pad weight test with vs without the pessary and/or >50% reduction in the average daily reports of number of urine leaks per day during periods with and without the pessary.

SECONDARY OUTCOMES:
Change in Quality of Life as measured by the Incontinence Impact Questionnaire Short Form (IIQ-7) at baseline and at the end of the treatment phase. | 24 days
  The IIQ-7 assesses the psychosocial impact of urinary incontinence in women, specifically physical activity, travel, social relationships and emotional health.

CONTACTS AND LOCATIONS:
Overall Officials: Melody A Roberts, Principal Investigator — Liv Labs Inc.
Locations (3):
- United States (3):
  - Northwestern Medicine Urogynecology and Reconstructive Surgery, Chicago, Illinois
  - Northwestern Medicine Urogynecology and Reconstructive Surgery, Lake Forest, Illinois
  - The Ohio State University Medical Center (OSUMC), Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No